CLINICAL TRIAL: NCT03316638
Title: Phase I/II Open Label Dose Escalation and Dose Expansion Study of Intravenous Infusion of W0101, an Antibody-drug Conjugate, in Patients with Advanced or Metastatic Solid Tumors. International, Multicenter, Open Label Study
Brief Title: A Study of a New Investigational Medicinal Product to Treat Patients with Advanced or Metastatic Solid Tumors
Acronym: Ulysse
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: delay in participants recruitment in cohort A3 and IMP manufacturing issues
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: W00101IV101
Record Dates: First submitted 2017-09-28; First posted 2017-10-20 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2022-12

CONDITIONS: Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Intervention Model Description: 2 Cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- W0101 - Cohort A1 (Experimental): This is a 14 days treatment cycle cohort in a 2 weeks schedule
  Interventions: Drug: W0101 - Cohort A1
- W0101 - Cohort A2 (Experimental): This is a 21 days treatment cycle cohort in a 3 weeks schedule
  Interventions: Drug: W0101 - Cohort A2
- W0101 - Expansion Phase (Experimental): Will be initiated after completion of cohorts A1 and A2
  Interventions: Drug: W0101 - Expansion Phase

INTERVENTIONS:
Drug: W0101 - Cohort A1 — Administered once every 2 weeks
  Other Names: Dose escalation Phase
  Arms: W0101 - Cohort A1
Drug: W0101 - Cohort A2 — Administered every 3 weeks
  Other Names: Dose escalation Phase
  Arms: W0101 - Cohort A2
Drug: W0101 - Expansion Phase — Administered according to the recommended dose for expansion
  Other Names: Expansion Phase
  Arms: W0101 - Expansion Phase

SUMMARY:
W0101 combines a cytotoxic compound to a monoclonal antibody targeting a receptor commonly overexpressed in many cancers.

The development of antibody-drug conjugates takes advantage of the specificity of the mAb while augmenting its ability to produce a cytotoxic effect. The expected benefits of antibody-drug conjugation are enhancement of cytotoxicity in target cells and limiting toxicities of cytotoxic drugs in normal tissues.

DETAILED DESCRIPTION:
This is a First In Human study, multicenter, open label study divided into 2 parts: an initial dose escalation phase (I) followed by expansion cohort(s) phase (II).

ELIGIBILITY:
Inclusion Criteria:

Dose escalation phase (cohort A1 and A2)

1. Male or female subjects age ≥ 18 years
2. Subjects with histologically or cytologically confirmed advanced or metastatic solid tumors (excluding lymphoma) , unresponsive to standard treatment or for whom no standard treatment is available or appropriate
3. ECOG performance status 0 or 1
4. Adequate bone marrow, renal, hepatic at screening and at Baseline
5. Subject must have measurable diseases as per RECIST v1.1 criteria

Exclusion Criteria:

1. Symptomatic brain metastases, CNS tumors
2. Symptomatic motor or sensory peripheral neuropathy (≥ grade 2)
3. Subjects having ophthalmologic abnormalities
4. Active serious systemic disease (infection,organic or dysmetabolic desease)
5. Left ventricular ejection fraction (LVEF) < 45% as determined by MUGA scan or echography at screening
6. QTc > 470 msec on screening ECG or congenital long QT syndrome
7. Biologic therapy (including ADCs ≤ 4 weeks before first study treatment administration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Specific Adverse Events | 28 days
  Identification of Dose-limiting toxicities
Incidence of Specific Adverse Events | From first administration up to 63 days
  Identification of Dose-limiting toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chetaille, MD, Study Chair — Pierre Fabre Medicament
Locations (3):
- France (2):
  - IUCT, Toulouse
  - IGR, Villejuif
- VHIO, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Undecided